CLINICAL TRIAL: NCT05818774
Title: A Prospective, Randomized, Double Blind Clinical Trial Comparing End-on Versus Parallel Radiofrequency Lesioning for Neurotomy of the Cervical Medial Branch Nerves: The EndPaRL Study
Brief Title: End-on Versus Parallel Radiofrequency Lesioning for Neurotomy of the Cervical Medial Branch Nerves
Acronym: EndPaRL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anuj Bhatia, Professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-5634
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain; Zygapophyseal Joint Arthritis
Keywords: Radiofrequency neurotomy; Cervical Medial Branch Nerves
MeSH Terms: conditions — Neck Pain | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFN of CMBNn with end-on lesioning with multitIned trident cannulae (Experimental): Intervention type: RF nerve end-on lesioning at 80-850 Celsius for 90 seconds
  Intervention name: End-on placement of the multitined trident cannulae
  Intervention description:
  Patient in lateral position, targeting joint position between the inferior C2 and superior C3 facets, the middle of the facet pillars for the third to fifth cervical levels, and the superior part of the sixth and seventh cervical facets
  Interventions: Procedure: Radiofrequency neurotomy (RFN) of Cervical Medial Branch Nerves (CMBNn) with end-on lesioning with multitined trident cannulae
- RFN of CMBNn with parallel lesioning with sharp straight conventional cannulae (SIS's technique) (Active Comparator): Intervention type: RF nerve parallel lesioning at 80-850 Celsius for 90 seconds
  Intervention name: Straight sharp conventional (SIS's technique)
  Intervention description:
  Technique as described in the SIS Practice Guidelines for parallel lesioning cannulae placement
  Interventions: Procedure: Radiofrequency neurotomy (RFN) of Cervical Medial Branch Nerves (CMBNn) with parallel lesioning

INTERVENTIONS:
Procedure: Radiofrequency neurotomy (RFN) of Cervical Medial Branch Nerves (CMBNn) with parallel lesioning — Intervention type: RF nerve lesioning at 80-85 degree Celsius for 90 seconds Intervention name: Straight sharp conventional (SIS's technique)
  Intervention description:
  Technique as described in the SIS Practice Guidelines for parallel lesioning cannulae placement
  Arms: RFN of CMBNn with parallel lesioning with sharp straight conventional cannulae (SIS's technique)
Procedure: Radiofrequency neurotomy (RFN) of Cervical Medial Branch Nerves (CMBNn) with end-on lesioning with multitined trident cannulae — Intervention type: RF nerve lesioning lesioning at 80-850 Celsius for 90 seconds Intervention name: End-on placement of the multitined trident cannulae
  Intervention description:
  Patient in lateral position, targeting joint position between the inferior C2 and superior C3 facets, the middle of the facet pillars for the third to fifth cervical levels, and the superior part of the sixth and seventh cervical facets.
  Arms: RFN of CMBNn with end-on lesioning with multitIned trident cannulae

SUMMARY:
Aim of the EndPaRL study is to compare the efficacy and effectiveness of the two techniques utilizing sharp straight conventional radiofrequency needle with a trident needle for radiofrequency neurotomy of Cervical Medial Branch Nerves (CMBNs), in patients presenting with chronic, moderate-to-severe, neck pain due to cervical zygapophyseal joint osteoarthritis, as diagnosed by positive responses to two consecutive diagnostic blocks with local anesthetic of the CMBN.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient of either gender aged 18-85 years
2. Predominant axial (non-radicular) neck pain for at least 3 months
3. 7-day average NRS score for neck pain ≥ 5/10 at baseline evaluation
4. Moderate or greater functional impairment due to pain, defined as NDI Questionnaire raw score of 15 out of 50 (≥30% )e Failure to respond to conservative medical management (pharmacologic, physical therapy) for at least 3 months;

f) Positive response to two consecutive diagnostic blocks of the CMBN with a short and long-acting anesthetic

Exclusion Criteria:

1. Participants with financial incentives or litigation associated with ongoing pain
2. Inability to complete assessment instruments
3. Chronic widespread pain
4. Prior RFN of the CMBN;
5. Severe mental health issues
6. Pregnancy or other reason that precludes the use of fluoroscopy
7. Untreated coagulopathy
8. Systemic or local infection at the time of screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Difference in mean Numerical Rating Scale (NRS) for pain scores | 3 months
  Difference in the mean pain scores before and after procedure. Scale from 0 to 10, where higher scores mean worse outcome
Proportion of patients with positive analgesic response | 3 months
  Proportion of patients with positive analgesic response (≥50% reduction in the NRS score for neck pain compared to baseline)

SECONDARY OUTCOMES:
Difference in the mean Numerical Rating Scale (NRS) for pain scores | at 1, 6 and 12 months
  Difference in mean NRS for pain scores at 1, 6 and 12 months after the RFA procedure. Scale from 0 to 10, where higher scores mean worse outcome
Proportion of patients with positive analgesic response | at 1,3, 6 and 12 months
  Proportion of patients with positive analgesic response (≥50% reduction in the NRS score for neck pain compared to baseline) at 1,3, 6 & 12 months
Proportion of patients with reduction in the Neck Disability Index (NDI) score | at 1, 3, 6, and 12 months
  Proportion of patients with ≥10% reduction in the NDI score at 1, 3, 6, and 12 months. Scale from 0 to 50, where higher scores mean worse outcome
Proportion of participants reporting improvement in the Patient Global Impression of Change (PGIC) scale | at 1, 3, 6, and 12 months
  PGIC score is a 7 point scale depicting a patient's subjective rating of overall improvement over time, as proportion of participants reporting improvement in the PGIC scale at 1, 3, 6, and 12 months
Difference in mean Pittsburgh Sleep Quality Index (PSQI) scores for sleep quality | at 1, 3, 6, and 12 months
  Difference in mean PSQI scores scores at 1, 3, 6, and 12 months. It has a range of 0-21; higher scores indicate worse sleep quality.
Difference in mean European Quality of Life (EQ-5D-5L score), a self-assessed, health related, quality of life questionnaire. It ranges from 5 to 25, where higher scores indicate worse outcome. | at 1, 3, 6, and 12 months
  Difference in mean EQ-5D-5L scores at 3, 6, and 12 months
Differences in duration of procedure between 2 groups | day of procedure
  Differences in duration of procedure in two groups
Differences in discomfort procedure between 2 groups | day of procedure
  Differences in patient discomfort of procedure
Differences in radiation dose of procedure between 2 groups | day of procedure
  Differences in radiation dose of procedure
Differences in cost of procedure between 2 groups | day of procedure
  Differences in cost of the procedures
Difference in opioid requirements in daily oral morphine equivalents between the groups | at 3, 6, and 12 months follow-ups after the procedure
  Difference in opioid requirements in daily oral morphine equivalents in mg averaged over the 1 week before and at 3, 6, and 12 months follow-ups after the procedure
Difference in average physical activity and sleep duration | 1 week before the procedure and 1 month after the procedure
  Difference in average physical activity and sleep duration as measured by wrist-worn actigraphy worn for 1 week before the procedure and 1 month after the procedure
Difference in incidence of peri-procedural complications and post-procedural adverse effects following the RFN procedure | at 1, 3, 6, and 12 months after the procedures
  Difference in incidence of peri-procedural complications and post-procedural adverse effects following the RFN procedure in the two groups during and at 1, 3, 6, and 12 months after the procedures
Patient assumption of the group assigned | at 3 months after procedure
  Patient assumption of the group assigned at 3 months after the RFN procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD, PhD, Principal Investigator — Department of Anesthesia and Pain Management, University Health Network, Toronto
Locations (3):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - University Health Network (UHN), Toronto, Ontario
- Division of Pain Medicine, Department of Anesthesiology, Reanimation, and Pain Medicine, Hospital Clínic de Barcelona, University of Barcelona., Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD at the moment

REFERENCES:
- [Background] MacVicar J, Borowczyk JM, MacVicar AM, Loughnan BM, Bogduk N. Cervical medial branch radiofrequency neurotomy in New Zealand. Pain Med. 2012 May;13(5):647-54. doi: 10.1111/j.1526-4637.2012.01351.x. Epub 2012 Mar 28. PMID 22458772
- [Result] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Result] Barnsley L. Percutaneous radiofrequency neurotomy for chronic neck pain: outcomes in a series of consecutive patients. Pain Med. 2005 Jul-Aug;6(4):282-6. doi: 10.1111/j.1526-4637.2005.00047.x. PMID 16083457
- [Derived] Alomari A, Ferreira-Dos-Santos G, Singh M, Burnham T, Cao X, McCormick Z, Flamer D, Kumar P, Hoydonckx Y, Khan JS, Tumber PS, Alvares D, Bhatia A. End-on versus parallel radiofrequency lesioning for neurotomy of the cervical medial branch nerves: a study protocol of a prospective, randomized, double-blind clinical trial: the "EndPaRL" study. Trials. 2023 Nov 11;24(1):721. doi: 10.1186/s13063-023-07752-9. PMID 37951900